CLINICAL TRIAL: NCT05918783
Title: A Multicenter Open-label Phase 1/1b Study to Evaluate Safety, Feasibility and Early Treatment Effect of Padeliporfin VTP Using Robotic Assisted Bronchoscopy and Cone Beam CT Guidance in Patients With Peripheral Lung Cancer
Brief Title: Padeliporfin VTP Using Robotic Assisted Bronchoscopy in Peripheral Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2201 LCM101
Record Dates: First submitted 2023-04-25; First posted 2023-06-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Lung Tumor
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Part B recruitment will be opened upon completion of Part A light dose escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Part A (Experimental): will be a monotherapy light dose escalation with single dose of Padeliporfin at light laser doses of 150, 250 and 400 mW/cm for 20 minutes.
  Part A will proceed with light dose escalation and will continue until the maximum tolerated light dose (MTD) and/or recommended phase 2 dose (RP2D) is defined.
  Interventions: Combination Product: Padeliporfin Vascular Targeted Photodynamic (VTP) therapy
- Part B (Experimental): will be a dose expansion part at MTD/RP2D dose level identified in Part A to further assess the safety, tolerability, and treatment effect of the MTD and/ or RP2D
  Interventions: Combination Product: Padeliporfin Vascular Targeted Photodynamic (VTP) therapy

INTERVENTIONS:
Combination Product: Padeliporfin Vascular Targeted Photodynamic (VTP) therapy — Bronchoscopy will be performed with robotic assisted approach using standard practices using general anaesthesia and placement of the optic fiber intratumorally followed by IV administration of Padeliporfin for 10 min and laser light illumination.
  Other Names: Padeliporfin VTP

SUMMARY:
Phase 1/1b, safety, feasibility, and light dose titration study followed by further study of therapeutic ablation effects.

Patients with high risk of peripheral primary lung cancer, stage 1A1/1A2, for whom surgical treatment is planned, will be recruited. Surgery will be performed at 5-21 days following the VTP procedure.

Study intervention: robotic assisted bronchoscopic Padeliporfin VTP lung ablation: vascular targeted photodynamic therapy using Padeliporfin photosensitizer.

DETAILED DESCRIPTION:
A multicenter, open label, phase 1/1b, safety, feasibility, and light dose titration study followed by further study of therapeutic ablation effects.

Patients with high risk of peripheral primary lung cancer, stage 1A1/1A2, for whom surgical treatment is planned, will be recruited. Patients who are candidates for lung resection will be recruited as a diagnose and treat in the same anaesthesia, protocol; surgery will be performed at least 5 days and up to 21 days following the VTP procedure.

Study intervention will consist of robotic assisted bronchoscopic Padeliporfin VTP lung ablation: vascular targeted photodynamic therapy using Padeliporfin photosensitizer, an ablation mechanism with efficacy related to immune response post-ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Patients with primary lung lesions who are at high risk for primary lung cancer.

   2.1.Biopsy with intraoperative confirmation of malignancy using on-site cytology will be used as final inclusion prior to study treatment.
3. All patients will be approved by a multi-disciplinary team (thoracic surgery, interventional pulmonology, medical oncology and radiation oncology) as appropriate for bronchoscopic VTP prior to surgical resection.
4. Tumor size targeted for VTP treatment ≤ 2 cm (Part A) and <3cm (Part B), based on CT scan, including solid or semi-solid tumors.
5. EBUS mediastinal staging performed intraoperative prior to VTP treatment with rapid on-site evaluation negative for nodal involvement of malignancy.
6. Tumor is ≥ 2cm from the central bronchial tree (distal 2 cm of the trachea, carina, and named major lobar bronchi up to their first bifurcation) (Timmerman, 2018).
7. Lung lesion is not contiguous with and ≥ 1 cm from the pleura/fissures.
8. Patient is eligible to undergo bronchoscopy under general anesthesia.
9. Tumor is accessible for Padeliporfin VTP treatment via robotic bronchoscopy
10. ECOG performance score 0-2
11. Estimated life expectancy of ≥3 months
12. Adequate organ system function
13. Negative serum pregnancy test

Exclusion Criteria:

1. Patient has a centrally located lung lesion, as defined by RTOG within 2 cm of the proximal bronchial tree, or within 2 cm of other major mediastinal structure (aorta, heart, trachea, pericardium, superior vena cava, pulmonary artery, esophagus, vertebra's body or spinal canal).
2. Patient has a lung lesion located less than 1 cm from the pleura or fissure
3. Patient has a lung cancer lesion >2cm in diameter, for the expansion cohort lesion >2-3 cm
4. Patient has cytologic or histologic evidence of nodal disease
5. Tumor invades major vessels
6. Prior exposure to VTP or PDT treatments
7. Pregnant or breastfeeding women
8. Receiving any other investigational treatment
9. Co-morbidities:

   1. Baseline hypoxia with O2 saturation <92% on 2L NC or more of oxygen
   2. New York Heart Association (NYHA) stage III/IV heart failure
   3. Unstable coronary artery disease or MI within the last 6 months
   4. Uncontrollable clinically serious arrhythmia
   5. Decompensated/clinically worsening interstitial lung disease or obstructive lung disease.
   6. Unstable cerebrovascular or peripheral vascular disease
   7. Inability to stop anticoagulation or anti-platelet therapy peri-procedure
   8. Evidence of clinically active infection requiring systemic (any route) antibiotic therapy. All prior infections must have resolved following optimal therapy.
   9. Patient has any acute or chronic condition assessed as clinically significant by Investigator which may preclude bronchoscopy procedure
   10. History of medical or psychiatric disease which, in the view of the investigator, would preclude safe treatment or acceptable study compliance
   11. Known severe pulmonary hypertension (mean pulmonary arterial pressure ≥ 50 mmHg)
10. Patient has a cancer diagnosis with active disease requiring further cancer therapy.
11. Patient has had major surgery within the last 4 weeks.
12. Patient has porphyria or hypersensitivity to padeliporfin or porphyrin-like compounds or to any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of robotic assisted bronchoscopic Padeliporfin VTP ablation | Day 30
  Incidence of treatment-related adverse events as assessed by CTCAE v5.0
Feasibility of robotic assisted bronchoscopic Padeliporfin VTP treatment | Day 1
  Feasibility of robotic bronchoscopic light fiber delivery into the target lesion as confirmed by cone beam CT and complete VTP treatment
Evaluate Maximum Tolerated light Dose and/or RP2D of Padeliporfin VTP ablation | Day 14
  Evaluate Maximum Tolerated light Dose and/or RP2D of robotic assisted bronchoscopic Padeliporfin VTP ablation (a vascular targeted photodynamic therapy with Padeliporfin of patients with peripheral stage 1A1/1A2) primary non-small cell lung cancers.

SECONDARY OUTCOMES:
Evaluation lung surgery feasibility | Day 5-21
  Number and severity of operative, postoperative adverse events Number and length of any delays to surgery or surgical cancellations Number of completed surgeries
Evaluation of the ablation area | 2 days post Padeliprofin VTP
  Acute radiographic changes on CT chest imaging obtained two days post Padeliporin VTP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No